CLINICAL TRIAL: NCT06155344
Title: VEGALIM : Vegetalization of the Maternal Diet During Pregnancy: Association With Pregnancy Outcomes and Newborn Health.
Brief Title: Vegetalization of the Maternal Diet During Pregnancy: Association With Pregnancy Outcomes and Newborn Health.
Acronym: VEGALIM
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: UMR 1280 PHAN (Unknown); INRAE - CRESS (Unknown)
Responsible Party: Sponsor
Other Study IDs: RC23_0399; 2023-A01997-38 (Other: ANSM)
Record Dates: First submitted 2023-11-06; First posted 2023-12-04 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Diet During Pregnancy
Keywords: Pregnancy; Newborn; Vegetalization; Food

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — One tube collection of 4 mL maternal blood in the first trimester and at delivery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women included in the VEGALIM project: Pregnant women consulting CEMAFOER (Center for Maternal and Fetal Pathology Screening and Risk Assessment) of Nantes University Hospital for pregnancy monitoring
  Interventions: Other: Food Frequency Questionnaire; Other: Collection of 4 mL maternal blood

INTERVENTIONS:
Other: Food Frequency Questionnaire — We will obtain a global index of vegetalization of the diet (the Plant based Diet Index: PDI) from data obtained using semi-quantitative questionnaires on food frequency (Food Frequency Questionnaire (FFQ)) validated on the national ELFE cohort (French Longitudinal Study from Childhood (https://www.elfe-france.fr)) and completed by women in the 1st trimester of pregnancy (T1) and at delivery.
Other: Collection of 4 mL maternal blood — One tube collection of 4 mL maternal blood in the first trimester and at delivery.

SUMMARY:
Reducing consumption of foods of animal origin in favor of more plant-based diets is a major environmental, public health and economic challenge. Data on the health effects of highly vegetalized diets are available only in adults. Few studies report the effect of the level of vegetalization of the maternal diet during pregnancy on the mother's health, and the development and health of the child. The VEGALIM project aims to describe the level of vegetalization of pregnant women's diets and the nutritional quality of their diets early in pregnancy (first trimester) and late pregnancy, and to explore the potential effects on their plasma lipid profile that may impact on their health during pregnancy and the health of the newborn.

ELIGIBILITY:
Inclusion Criteria :

* Pregnant women consulting the CEMAFOER at the Nantes University Hospital for pregnancy monitoring
* Gestational age between 11 and 13 AW +6 days
* Understanding French

Exclusion Criteria:

* Patients under 18 years of age
* Patient who objected to being included in the study
* Patient with cognitive problems that prevent her from answering questionnaires

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be included during the 1st trimester follow-up visit (at 11-13 amenorrhea weeks (AW) + 6 days), organized by the maternal and fetal pathology screening and risk assessment center (CEMAFOER) at the Nantes University Hospital. Patients will then be informed of the research project, and their written consent to participate in the study will be obtained.
Sampling Method: Non-Probability Sample
Enrollment: 670 (Estimated)
Dates: Start 2024-03-18 (Actual); Primary Completion 2027-06-18 (Estimated); Study Completion 2027-12-18 (Estimated)

PRIMARY OUTCOMES:
Characterizing the levels of plant-based food consumption at the beginning of pregnancy (at the end of the first trimester of pregnancy) based on the completion of the Food Frequency Questionnaire (FFQ, scale from 0 to 6 ; 0 being the worst outcome) | 25 minutes

SECONDARY OUTCOMES:
Study the evolution of the vegetation score between the 1st and 3rd trimester of pregnancy | 6 months
Study changes in diet quality between the 1st and 3rd trimesters of pregnancy | 6 months
Studying the association between vegetarian diets in the first trimester of pregnancy and pregnancy outcomes (such as prematurity, birth weight, maternal pathologies not present at the time of inclusion (gestational diabetes, pre-eclampsia, etc.). | 6 months
Study the association between diet quality in the first trimester of pregnancy and pregnancy outcomes (such as prematurity, birth weight, maternal pathologies not present at the time of inclusion (gestational diabetes, pre-eclampsia, etc.). | 6 months
Study the association between the vegetalization of the diet and the lipid profile of women in the 1st trimester and at childbirth. | 6 months
Study the association between diet quality and lipid profiles of women in the 1st trimester and at childbirth. | 6 months
Study the association between the vegetalization of the diet and the total fatty acid status of women in the 1st trimester and at childbirth. | 6 months
Study the association between diet quality and total fatty acid status in women at 1st trimester and at childbirth. | 6 months
Identify other biological markers, such as vitamins, that may be impacted by a change in diet, and study the influence of diet quality on these potential plasma markers of patient and of Umbilical cord blood plasma. | 6 months
Study the association between diet quality and the lipid profile of umbilical cord blood at delivery (T3). | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Winer, MD, PHD, Principal Investigator — Nantes University Hospital; Veronique Ferchaud-Roucher, PhD, Study Director — UMR 1280 PHAN
Locations (1):
- CHU de Nantes, Nantes, Loire-Atlantique, France

IPD SHARING:
Plan to Share IPD: Undecided